CLINICAL TRIAL: NCT01301235
Title: Defining 31Phosphorous Magnetic Resonance Spectroscopy Characteristics of the Vastus Lateralis After Sub-maximal Exercise in Patients With Mitochondrial Myopathy
Brief Title: Defining 31Phosphorous Magnetic Resonance Spectroscopy Characteristics in Patients With Mitochondrial Myopathy
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Amy Fleischman, MD, Clinical Investigator, Massachusetts General Hospital
Other Study IDs: 2010P002441
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Mitochondrial Disease
Keywords: Mitochondria
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with mitochondrial disease

SUMMARY:
This is a developmental protocol to determine the MRI based 31P-MRS changes seen in subjects with mitochondrial myopathy using our dynamic exercise protocol and to identify the ideal variable(s) to represent mitochondrial function.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ age 18 years old with primary mitochondrial myopathy
2. Known alteration in electron transport chain activity (<25 % activity of ETC) or known mutations in mitochondrial gene.

Exclusion Criteria:

Failure based on standard clinical MRI Screening form - the form is intended to establish the safety of subjects participating in the MRI scan without divulging any confidentiality information -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with mitochondrial disease
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
PCr recovery after submaximal exercise by 31P-MRS | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States